CLINICAL TRIAL: NCT06568107
Title: A Person-Centered Environmental and Sensory Intervention for Nursing Home Residents With Dementia Who Exhibit Persistent Vocalizations
Brief Title: Environmental and Sensory Intervention for Nursing Home Residents With Dementia Who Exhibit Persistent Vocalizations
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2003007693; 5K23NR018673 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Environment; methyl hydroxyethyl cellulose; Methods

STUDY DESIGN:
Intervention Model Description: Single group - all participants enrolled in the study will receive the non-pharmacological intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EASE Intervention (Experimental): Thirty-two persons with dementia will be exposed by an interventionist to an Environmental And Sensory Experience (EASE) intervention which involves a tailored, person-centered nature scene projected with associated nature sounds. A within-person design will be used where the participants will serve as their own controls and be observed 30 minutes prior to, 30 minutes during, and for 30 minutes directly after EASE.
  Interventions: Behavioral: Environmental And Sensory Experience (EASE) intervention

INTERVENTIONS:
Behavioral: Environmental And Sensory Experience (EASE) intervention — The participant will be exposed to 30 minutes of a still nature image and associated nature sounds (60-80 beats per minute). An brief interview will occur with the legally authorized representative to find out what nature scene would meet the preference of the person living with dementia and persistent vocalizations.

SUMMARY:
The purpose of this study is to test a person-centered, nature-based non-pharmacological intervention for nursing home residents living with dementia who exhibit persistent vocalizations. The Environmental And Sensory Experience (EASE) involves the projection of a still nature image and the playing of nature sounds. Family members of the person living with dementia provide consent for the resident to participate in the study and complete a brief survey on nature preferences on the resident's behalf. The survey informs the research team on what nature scene to show. Participants will wear a watch that measures stress levels and research staff will monitor vocalization patterns. We will also recruit persons living with dementia from other settings such as assisted living, personal care units, and adult day care settings.

DETAILED DESCRIPTION:
After enrolling in the study, participants will participate in three study visits. During the first two visits, study personnel will observe the nursing home resident to collect data on the resident's vocalizing behaviors (persistent vocalizations, PVs). These visits will last for roughly six hours, one during the day shift and one during the evening shift. The third visit will last approximately 90 minutes. During this visit, study personnel will observe vocalizing behaviors before, during, and after the EASE intervention is in use. Residents will also wear a watch for all three visits that records information about their heart rate and stress levels. All visits will occur in the resident's natural environment- either their room or common space and will be scheduled at the convenience of the resident and NH staff.

The aims of the study are:

Aim 1: Examine the feasibility and preliminary efficacy of the EASE to reduce PVs among NH residents.

Aim 2: Evaluate the NH staff perception of the acceptability of the EASE within 48 hours post-intervention.

Aim 3: Examine the mechanism of action of the EASE.

ELIGIBILITY:
Inclusion Criteria:

* The participants must: 1) have a medical diagnosis of dementia; 2) have severe dementia as determined by a MMSE score of ≤9 (or another cognitive test indicating severe dementia); 3) have a history of PVs per staff report; 4) be 50 years older or greater; 5) require extensive assistance by staff to ambulate or is non-ambulatory (to allow for consistent video recording). In addition, consent will be obtained from the resident's Legally Authorized Representative (LAR) and assent from the participant.

Exclusion Criteria:

* Persons living with dementia will be excluded if they: 1) are blind; 2) are deaf; 3) give indications of dissent. Variations will be sought for gender, race and ethnicity.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Persistent Vocalizations (PVs) | 90 minutes
  Persistent vocalization (PV) duration will be recorded for the 90 minutes (prior to-, during-, and immediately after the EASE), and calculated for the 30 minutes prior to the intervention, the 30 minutes during the intervention, and 30 minutes immediately following the intervention. The interventionist will be video recording the participant only during the 90-minute observation time period. Digital video recording in this study will allow for quantifying start and stop times of the PVs to measure frequency and duration of PVs. A PV will be considered ended once it had stopped for 5 seconds. Duration of PVs will be tracked real-time on a paper form if the legally authorized representative opts out of video recording. A decline to video record option is present on the informed consent form, and if selected will not exclude participant. Analysis will involve looking at the duration and frequency of PVs during the 3- time points.

SECONDARY OUTCOMES:
Heart Rate (HR) | 90 minutes
  Heart rate will be collected via a wrist sensor 30 minutes prior to the intervention, the 30 minutes during the intervention, and 30 minutes immediately following the intervention. Analysis will include looking at heart rates during the 3-time points.
Electrodermal Activity | 90 minutes
  Electrodermal activity will be collected via a wrist sensor 30 minutes prior to the intervention, the 30 minutes during the intervention, and 30 minutes immediately following the intervention. Analysis will include looking at heart rates during the 3-time points.
Acceptability of Intervention Measure | 5 minutes
  This structured survey poses 4 statements, allows for customization to insert intervention name, and has the respondents use a 5-point Likert from completely disagree to completely agree. The statements are: 1) the EASE meets my approval, 2) the EASE is appealing to me, 3) I like EASE, and 4) I welcome EASE. Stakeholder NH staff (Nurses, Nursing Assistants and Administrators) working on the unit the participants live on will we be asked these questions with 48 hours following the intervention delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Justine S Sefcik, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No